CLINICAL TRIAL: NCT06099951
Title: Single Arm Phase II Clinical Trial of Recombinant Humanized Anti PD-1 Monoclonal Antibody and FOLFOXIRI Regimen Combined With Preoperative Intensity Modulated Radiation Therapy as the Total Neoadjuvant Treatment for pMMR Locally Advanced Low Rectal Cancer
Brief Title: Total Neoadjuvant Treatment for pMMR Locally Advanced Low Rectal Cancer: Anti-PD-1 Antibody With FOLFOXIRI and Preoperative Radiation Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHI-ZHONG PAN, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-173-Department of CRC
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Neoadjuvant chemoradiotherapy; Neoadjuvant immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Serplulimab+FOLFOXIRI (Experimental)
  Interventions: Drug: Serplulimab + FOLFOXIRI; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Serplulimab + FOLFOXIRI — Starting from day 0, the patient will receive 8 cycles of FOLFOXIRI regimen at specific intervals. The FOLFOXIRI regimen includes irinotecan 165mg/m2, oxaliplatin 85mg/m2, calcium folinate 200mg/m2 on day 1, followed by continuous intravenous infusion of 5-FU 2400mg/m2/day for 46 hours. This regimen is repeated every 14 days.During radiotherapy (Monday to Friday), the patient will receive capecitabine 1650mg/m2/day orally twice daily. Serplulimab immunotherapy will be administered every 2 weeks during the FOLFOXIRI neoadjuvant chemotherapy period. Serplulimab will be given on the first day and the 14th day of radiotherapy, dissolved in 100ml normal saline and administered intravenously over 30-60 minutes at a dose of 200mg.
Radiation: Radiation therapy — Radiation therapy

SUMMARY:
For locally advanced rectal cancer, the initial goal of neoadjuvant chemoradiotherapy is to reduce local recurrence, but the pathologic complete response (PCR) rate is low, and distant metastasis becomes the main treatment failure pattern. With the gradual optimization of neoadjuvant chemotherapy regimens, the tumor regression efficacy in patients has improved, leading to increased organ preservation and reduced distant metastasis. Therefore, neoadjuvant treatment for locally advanced rectal cancer has transitioned from an era focused on local control of recurrence to an era focused on improving tumor regression, organ preservation, and long-term survival. Thus, there is a trend towards intensifying the whole course of neoadjuvant treatment for rectal cancer to preserve organ function. The combination of chemotherapy, immunotherapy, and radiotherapy is currently the most powerful approach to maximize tumor regression and achieve organ preservation in low rectal cancer. Currently, several clinical studies on the use of PD-1 inhibitors in combination with preoperative chemoradiotherapy for locally advanced rectal cancer are ongoing internationally, with the majority focusing on PD-1 monotherapy or PD-1 combined with the CapOX regimen in combination with synchronous chemoradiotherapy as neoadjuvant treatment. However, there is no specific research reported on the use of PD-1 combined with FOLFOXIRI regimen in combination with synchronous chemoradiotherapy as a whole course neoadjuvant treatment for pMMR (proficient mismatch repair) locally advanced rectal cancer. Based on the above evidence from evidence-based medicine, we plan to conduct a phase II prospective clinical study to explore the efficacy and treatment safety of PD-1 monoclonal antibody and FOLFOXIRI chemotherapy combined with intensity-modulated radiotherapy as a whole course neoadjuvant treatment in pMMR locally advanced low rectal cancer. The results of this study may open up new treatment approaches for optimizing whole course neoadjuvant chemotherapy in locally advanced rectal cancer and provide a novel treatment strategy for organ preservation in pMMR rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* The pathological confirmation is rectal adenocarcinoma. Additionally, the tumor biopsy immunohistochemistry indicates pMMR, with all MSH1, MSH2, MSH6, and PMS2 showing positive expression.
* Age: 18 to 75 years old,allgenders
* MRI examination confirms that the lower margin of the tumor is within 5cm from the anal verge.
* Clinical stage cT3-4N0M0 or cTxN+M0, with or without positive MRF, with or without positive EMVI, estimated to be eligible for R0 resection.
* No signs of intestinal obstruction before surgery; or resolution of obstruction after proximal colostomy surgery
* Performance status (ECOG score) ≤ 2
* Hematology: WBC > 3 × 10^9 / L; PLT > 80 × 10^9 / L; Hb > 90 g/L;
* Liver function: ALT and AST ≤ 2.5 × ULN; bilirubin ≤ 1.5 × ULN;
* Renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CCr) ≥ 60 ml/min;
* Signed informed consent, willingness to undergo treatment according to this protocol, and good compliance with medication.
* No history of prior surgery, chemotherapy, radiation therapy, or immunotherapy.

Exclusion Criteria:

* Co-existing with other serious illnesses, including severe electrolyte disorders, bleeding tendencies, etc.
* Active or uncontrolled severe infections: a) Known human immunodeficiency virus (HIV) infection. b) Known clinically significant liver disease history, including viral hepatitis [known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e., HBV DNA positive (>1×104 copies/mL or >2000 IU/mL)]. c) Known hepatitis C virus (HCV) infection with positive HCV RNA (>1×103 copies/mL), or other hepatitis, liver cirrhosis.
* Women who are pregnant or breastfeeding and have childbearing potential but are not taking adequate contraceptive measures.
* Patients with severe brain disorders or mental illnesses (such as depression, mania, obsessive-compulsive disorder, and schizophrenia) that affect the patient's ability to self-report.
* Patients with autoimmune diseases, blood system disorders, and a history of organ transplantation, long-term use of steroids, or immunosuppressive agents
* History of other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ or basal cell carcinoma of the skin.
* History of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation).
* Hypertension that cannot be well controlled with antihypertensive medications (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete tumor response rate. | Immediately After obtaining the surgical specimen.
  Including pathological complete response (pCR) and clinical complete response (cCR); pathological complete response is defined as the absence of visible tumor cells in the rectal specimen obtained during surgery

SECONDARY OUTCOMES:
Sphincter preservation rate | During surgery
  Rate of patients preserving the anal sphincter during surgery

IPD SHARING:
Plan to Share IPD: No